CLINICAL TRIAL: NCT03380689
Title: Phase I Study of Combination Therapy With S-1, Irinotecan, and Bevacizumab as 1-line Chemotherapy in Patients With Advanced Colorectal Cancer.
Brief Title: Phase I Study of Biweekly SIRB Regimen for Metastatic Colorectal Cancer
Acronym: SIRB2
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: There is no fund to support it
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FNF008
Record Dates: First submitted 2017-12-17; First posted 2017-12-21 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2017-12

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — S 1 (combination); Irinotecan; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIRB2 (Experimental): Biweekly combination therapy with S-1, Irinotecan, and Bevacizumab
  Interventions: Drug: S-1; Drug: Irinotecan; Drug: Bevacizumab

INTERVENTIONS:
Drug: S-1 — - S-1 is administered orally on days 1 to 7 of a 14-day cycle. Patients are assigned on the basis of body surface area (BSA) to receive one of the following oral doses twice daily: 40 mg (BSA <1.25m2), 50 mg (BSA >1.25 to <1.50 m2), or 60 mg (BSA >1.50 m2).
  Other Names: S1
Drug: Irinotecan — - CPT-11 was administrated as a 90-min intravenous infusion on day 1 of a 14-day cycle. Five escalating dose levels of CPT-11 were prepared, at an initial dose of 75mg/m2/day (level 1), stepping up to 100 (level 2), 125 (level 3), 150 (level 4) or 175 (level 5) mg/m2/day.
  Other Names: CPT-11
Drug: Bevacizumab — - Bevacizumab (5 mg/kg) is administered by intravenous infusion over the course of 30 to 90 min on day 1 of each 2-week cycle.
  Other Names: Avastin

SUMMARY:
Phase I Study of biweekly combination therapy with S-1, Irinotecan, and Bevacizumab as 1-line Chemotherapy in Patients With Advanced Colorectal Cancer.

DETAILED DESCRIPTION:
In several clinical studies from Japan and South Korea, the combination regimen of S-1 and irinotecan has shown efficacy in the treatment of advanced colorectal cancer, and a Phase III study（TRICOLORE） showed that the combination therapy with S-1/irinotecan/bevacizumab (a 3-week regimen [SIRB] or 4-week regimen [IRIS/bevacizumab]) is not inferior to the oxaliplatin-based standard treatment (mFOLFOX6/bevacizumab or CapeOX/bevacizumab) in patients with metastatic colorectal cancer who had not previously received chemotherapy. Here, we design this phase I study to explore the Chinese population's tolerability and efficacy of Biweekly SIRB Regimen(S-1/irinotecan/bevacizumab) and to explore the recommended dose of irinotecan in this regimen.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal carcinoma with inoperable, locally advanced, or metastatic disease, not amenable to curative therapy
* Measurable disease or non-measurable but assessable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST)
* Patients with no previous treatment (radiotherapy or chemotherapy). Patients who have received postoperative adjuvant chemotherapy are eligible if relapse is diagnosed more than 180 days after the end of such treatment.
* Age ≥20 years
* Life expectancy of at least 3 months
* ECOG PS of 0 or 1
* Adequate function of major organs as defined below:

  * Hemoglobin ≥9.0g/dL
  * White blood cell count ≥3,500/mm3
  * Neutrophil count ≥1,500/mm3
  * Platelet count ≥100,000/mm3
  * AST and ALT ≤100 U/L (<200 U/L in patients with liver metastasis)
  * Serum creatinine ≤1.2 mg/dL

    * Creatinine clearance estimate by the Cockcroft-Gault method >50 mL/min (reduce initial dosage by one step if ≥50 but <80 mL/min)
* Able to take capsules orally.
* No electrocardiographic abnormalities within 28 days before enrollment that would clinically preclude the execution of the study, as judged by the investigator.
* Voluntary written informed consent.

Exclusion Criteria:

* Serious drug hypersensitivity or a history of drug allergy
* Active double cancer
* Active infections (e.g., patients with pyrexia of 38℃ or higher)
* History of gastrointestinal perforation, intestinal tract paralysis, or ileus within 1 year.
* Uncontrolled hypertension
* Serious complications (e.g., pulmonary fibrosis, interstitial pneumonitis, heart failure, renal failure, hepatic failure, or poorly controlled diabetes)
* Moderate or severe ascites or pleural effusion requiring treatment
* Watery diarrhea
* Treatment with flucytosine or atazanavir sulfate
* Metastasis to the CNS
* Pregnant women, possibly pregnant women, women wishing to become pregnant, and nursing mothers. Men who are currently attempting to conceive children.
* Severe mental disorder
* Continuous treatment with steroids
* Urine dipstick for proteinuria should be <2+
* Patient with a past history of thrombosis, cerebral infarction, myocardial infarction, or pulmonary embolism
* Major surgical procedure, open biopsy, or clinically significant traumatic injury within 4 weeks
* Long-term daily treatment with aspirin (>325 mg/day)
* History or evidence of inherited bleeding diathesis or coagulopathy with the risk of bleeding
* Judged ineligible for participation in the study by the investigator for safety reasons.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-05 (Estimated); Primary Completion 2018-07-05 (Estimated); Study Completion 2019-01-05 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerance dose | From enrollment to completion of study. Estimated about 12 months.
  Maximum tolerance dose (MTD) is the dose of treatment in the cohort where there are 2 cases of DTL reported.

SECONDARY OUTCOMES:
Dose limiting toxicity | From enrollment to completion of study. Estimated about 12 months.
  Dose limiting toxicity (DLT) is referred to grade 3 non-hematological toxicity or grade 4 hematological toxicity according to NCI CTCAE 4.03 criteria.
Objective response rate | From enrollment to 6 months after treatment.
  Clinical response of treatment according to RESIST v1.1 criteria (ORR, objective response rate).
Progression-free survival | From enrollment to progression of disease. Estimated about 6 months.
  The length of time from enrollment until the time of progression of disease (PFS, progression-free survival).
Overall survival | From enrollment to death of patients. Estimated about 1 year.
  The length of time from enrollment until the time of death (OS, overall survival).

CONTACTS AND LOCATIONS:
Overall Officials: Rongbo Lin, MD, Study Chair — Fujian Cancer Hospital
Locations (1):
- Rongbo Lin, Fuzhou, Fujian, China